CLINICAL TRIAL: NCT01852500
Title: Are Newborns Conscious of the Placebo Effect? Result From an RCT in Osteopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: European Institute for Evidence Based Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEO-Plac 01; NEO-Plac 01 (Other: AIOT IRB)
Record Dates: First submitted 2013-05-09; First posted 2013-05-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Sham OMT (Experimental): patients under standard medical care plus sham OMT
  Interventions: Other: Sham Osteopathic Manipulative Treatment
- Control (Other): patients under standard medical care plus only osteopathic evaluation
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Sham Osteopathic Manipulative Treatment — Patients from this group received sham osteopathic treatments twice a week for the entire length of stay in the unit.
  Arms: Sham OMT
Other: Standard care — Patients from control group received standard care plus osteopathic evaluation only, according to the same schedule as the study group.
  Arms: Control

SUMMARY:
Results from previous studies suggest the association between Osteopathic Manipulative Treatment (OMT) and length of stay (LOS) reduction in a population of preterm infants.

The primary objective of the present study is to evaluate the effectiveness of sham OMT in reducing LOS in a sample of preterm newborns, in order to investigate whether previous clinical results could be related to a hypothetical placebo effect.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants born at age between 29 and 37 weeks
* sham osteopathic treatment performed < 14 days after birth
* preterm infants born in the same hospital

Exclusion Criteria:

* gestational age < 29, > 37 weeks;
* sham osteopathic treatment performed > 14 days after birth;
* newborn transferred to/from other hospital;
* newborn from to HIV seropositive and/or drug addict mother;
* newborn with genetic disorders, congenital abnormalities, cardiovascular abnormalities, neurological disorders, proven or suspected necrotizing enterocolitis with or without gastrointestinal perforation, proven or suspected abdominal obstruction, pre- and/or post-surgery patients, pneumoperitoneum and/or atelectasis.

Ages: 29 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of sham OMT in reducing LOS | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

SECONDARY OUTCOMES:
pre-post difference in weight gain | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cerritelli, DO, MS, Study Chair — European Institute for Evidence Based Osteopathic Medicine
Locations (1):
- Francesco Cerritelli, Pescara, PE, Italy

REFERENCES:
- [Background] Cerritelli F, Pizzolorusso G, Ciardelli F, La Mola E, Cozzolino V, Renzetti C, D'Incecco C, Fusilli P, Sabatino G, Barlafante G. Effect of osteopathic manipulative treatment on length of stay in a population of preterm infants: a randomized controlled trial. BMC Pediatr. 2013 Apr 26;13:65. doi: 10.1186/1471-2431-13-65. PMID 23622070
- [Background] Pizzolorusso G, Turi P, Barlafante G, Cerritelli F, Renzetti C, Cozzolino V, D'Orazio M, Fusilli P, Carinci F, D'Incecco C. Effect of osteopathic manipulative treatment on gastrointestinal function and length of stay of preterm infants: an exploratory study. Chiropr Man Therap. 2011 Jun 28;19(1):15. doi: 10.1186/2045-709X-19-15. PMID 21711535